CLINICAL TRIAL: NCT05614479
Title: Healthy Lifestyle Habits Promotion to Improve Elderly People Health
Brief Title: Health Promotion Community-based Intervention Among Elderly People Through Self-managed MAHA Mobile App.
Acronym: Gatekeeper
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosistemak Institute for Health Systems Research (Other)
Collaborators: Basque Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 857223
Record Dates: First submitted 2022-10-17; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy; Chronic Disease
Keywords: Health promotion; Community based intervention; Healthy habits; Healthy lifestyle; Wellbeing; Innovative solutions; Quality of life; Self-care; Maintaining functionality; Active ageing; Empowerement; Educative health materials; Health literacy; Socialization; Community; Ageing; Older people
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, longitudinal (pre-post, prospective and without a control group). This research is not a clinical trial, but a technology testing study at community level (community intervention). Therefore, the health and medical treatments provided to the person do not differ from those provided to the participants. Nevertheless, the participant is entitled to know of any unexpected discoveries or findings as part of research conducted in a study, just as if the individual were not participating in the study. The mixed-method approach will provide scientific evidence based on the effectiveness, and user experience of a self-managed mobile health application that recommends activities to promote healthy lifestyle habits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): Use of the MAHA mobile application
  Interventions: Other: GATEKEEPER intervention

INTERVENTIONS:
Other: GATEKEEPER intervention — Agents will identify candidates in their areas of work (e.g., associations of elderly people).
  Training sessions will be held for healthcare professionals and community agents.
  Dissemination of materials, resources, and channels to contact and inform candidates to invite them to participate in the study. Recruitment procedures posters, leaflets, videos, newsletters, or appointments will be used.
  Candidates interested and accepted will download the application on their mobile devices and will surf on the app which pretends to promote healthy aging. Users will provide some data and complete questionnaires (available in the application) for the baseline and final assessment.
  Professionals will visualize how and how much participants are interacting by using the MAHA dashboard.

SUMMARY:
The GATEKEEPER project, funded by the European Commission's HORIZON 2020 innovation framework, aims to ensure healthier independent living for ageing populations. To this end, GATEKEEPER aims to develop an open, European-wide, standards-based, interoperable and secure platform, available to all stakeholders (healthcare professionals, technology companies and users), offering digital solutions on the Internet of Things, Big Data or Artificial Intelligence, or new techniques, for early detection and personalised interventions to ensure healthier independent living for ageing populations.

GATEKEEPER will demonstrate its value by scaling up innovative solutions, during a 48-month work plan that will involve 40.000 elderly citizens, as well as authorities, institutions, companies, associations and academic centres from 8 pilot regions in 7 EU Member States. The pilots sites will deploy and demonstrate the effect, benefit, value and scalability of GATEKEEPER solutions around reference use cases covering primary, secondary and terciary prevention in the Basque Country (Spain), Aragon (Spain), Attica and Central Greece (Greece), Cyprus (Cyprus), Lodz (Poland), Milton Keynes (UK), Puglia (Italy) and Saxony (Germany).

The Basque Country pilot site is involved in the Reference Use Cases focused to "Lifestyle-related early detection". The intervention aims to encourage active and healthy ageing by the use of a self-managed mobile application, thereby to enhance independence, autonomy and improve the well-being of older people, promoting their physical, cognitive and mental activity and social participation. This quasi-experimental and longitudinal study is target to 10,000 older people and/or their caregivers from the Basque Country region. A multi-channel and community-based recruitment strategy at Basque regional level has been designed that involves 39 community-based organizations from the Basque Health Ecosystem.

DETAILED DESCRIPTION:
The population over 65 years of age in OECD (Organisation for Economic Co-operation and Development) countries has been increasing in recent years. In 2010 it was 15% and is expected to reach 22% by 2030. Life expectancy of people aged 65 has also increased significantly over the last 50 years, being higher in OECD countries, with women living 21 years longer and men 17 years longer, representing an increase of almost 40% since 1960. This demographic change of society in the European Union (EU) leads to increased costs in health and social care systems, as care and prevention measures for all ages are becoming increasingly expensive.

To tackle this challege, health systems should identify solutions that improve the lifelong health and well-being of elderly people, and hence the effectiveness of prevention, treatment and management of disease and disability.

The European funded GATEKEEPER project aims to ensure healthier independent living for ageing populations. As a result, GATEKEEPER will deploy an open, European-wide, standards-based, interoperable and secure platform, available to all stakeholders (healthcare professionals, technology companies and users), offering digital solutions on the Internet of Things, Big Data or Artificial Intelligence, or new techniques, for early detection and personalised interventions to ensure healthier independent living for ageing populations. The study will engage 40,000 senior citizens, as well as authorities, institutions, companies, associations and academic centres from 8 pilot regions in seven medical use cases.

The Basque Country region participates the "Lifestyle-related early detection" use case. It has implemented a health promotion intervention to encourage active and healthy ageing of Basque elderly people by the use of a self-managed MAHA mobile application. The main objective is to assess the effectiveness and user experience of a self-managed mobile health application that recommends activities to promote healthy lifestyle habits. Secondary objectives are:

* To encourage active and healthy ageing, promoting physical activity, cognitive training and social participation.
* To enhance independence, autonomy and improve the well-being of older people.
* To increase the empowerment of older people and their caregivers, family members or reference people.

This quasi-experimental and longitudinal study is aiming to target 10,000 older people and/or their caregivers from the Basque Country (Spain). Recruitment will follow a multi-channel and community based strategy at Basque regional level. More than 25 community based organizations from the Basque Health Ecosystem are participating in the intervention. The professionals as recruiters disseminate the intervention and invite participants who meet the inclusion criteria (people over 65 years old and/or caregivers that are familiar with mobile and technologies) to use the ehealth Appl for improving their health, daily habits and enhance health literacy.

The study will have a total duration of 24 months structures in three phases: intervention design and preparation; running phase, and evaluation process. In the 1st phase, the process of adapting and customising the technology to the needs of the study has been carried out. In parallel, professionals from key organizations at community setting has been invited to participate in the development, identification and review of the contents, usability and interface of the App mock-ups. In the 2nd phase, as part of the intervention running phase, traning sessions with healthcare professionals and community-based professionals have been carried out. Trained professionals through dissemination materials and channels (posters, explanatory leaflets, videos, newsletters or face-to-face appointments) start contacting and informing the study candidates to participate in the intervention. Candidates who are interest and accept to participate will download the application on their mobile devices and start using MAHA. The 3rd and last phase will conduct an evaluation where the intervention research question will be answered. The research question is: Can ehealth mobile application promote habits and attitudes that lead to healthy lifestyles, enchace independence, and autonomy and increase the empowerment among elderly people? The intervention aforementioned started in April 2022, once traning sessions with the profesionals at community-based organizations held. The project envisages between six and 9 month window from the start of the intervention to achieve the total number of citizen recruited. During the intervention period, citizen will use the MAHA App that will offer activities, materials and contents to reinforce the socialization, promote habits and attitudes that lead to healthy lifestyles, push active ageing and empowerment, and delay or reduce the deterioration of the health. The intervention will end in September 2023, after which the evaluation will be carried out to analyse if MAHA has contributed to make senior healthier and make healthy choices easier! A mixed methods approach will be employed, which refers to an emerging research methodology that advances the systematic integration of quantitative and qualitative data into a single investigation. Data collected from participants' MAHA application will be used for quantitative evaluation. It will be conducted a baseline assessment, by collecting the following questionnaires at baseline, one the participant has registered in the App: EuroQoL-5D and Get up from the chair 5 times test from the app server. The final evaluation will take place at the end of the defined monitoring period. This evaluation will be based on information from quantitative data collected through questionnaires (EuroQoL-5D, Get up from your chair 5 times test and MAUQ) and usage metrics from the app server.

Data management comply with the new EU regulation on data protection (General Data Protection Regulation, GDPR) that has entered into force on 28 May 2018. The GATEKEEPER I study will only collect essential data that will come from the app server (all data extracted from the app server and used for analysis will be anonymised) and information from focus groups and/or semi-structured interviews with professionals practitioners (data for analysis will be pseudonymised). This data processing will be carried out in accordance with the data protection regulation no. 2016/679. Only those responsible for the evaluation (Osakidetza-Basque Health Service) of the Basque Country team will have access to identifiable data in a protected environment. Those responsible for the evaluation will sign an express commitment to confidentiality and not to carry out any re-identification activity.

App user data transferred to the evaluation team (Open Evidence, the Gatekeeper partner responsible for the evaluation of the project) and usage metrics transferred to the Gatekeeper platform (hosted by the Universidad Politécnica de Madrid, a GATEKEEPER partner) will be anonymised. The data transfer mechanisms between European regions will comply with the new EU regulation on data protection (General Data Protection Regulation, GDPR) that has entered into force on 28 May 2018.

ELIGIBILITY:
PARTICIPANTS -Inclusion criteria

* Subjects are eligible for the study if they are:
* 65 years of age or older and/or their caregiver, family members and reference people
* With stable internet access and at least one of the following devices to use the GATEKEEPER application: Smartphone or Tablet
* They or their informal caregivers understand, read and talk the native language.

PARTICIPANTS -Exclusion criteria

Patients are not eligible for recruitment if:

* Aged < 65 years
* Do not have access to internet or at least one of the following devices to use the GATEKEEPER application: Smartphone or Tablet

INFORMAL CAREGIVERS- Inclusion criteria

The informal caregiver will be a person who provides occasional or regular support to the participant. Caregivers are eligible if:

* The participant they take care of meet the inclusion criteria
* They have stable internet access and at least one of the following devices to use the GATEKEEPER application: Smartphone or Tablet

INFORMAL CAREGIVERS-Exclusion criteria Caregivers are not eligible if the user meets the exclusion criteria.

PROFESSIONALS-Inclusion criteria

Professionals are eligible if they have a direct connection with participants who meet the inclusion criteria and accept to participate. Professionals taking part in GATEKEEPER intervention should be:

• open to the use of new technology. They should be willing to learn how to use technology to support users if needed.

PROFESSIONALS-Exclusion criteria Professionals are not eligible if they do not care for users who meets the inclusion criteria or only care for patients who meet the exclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of Life by EuroQoL-5D | Change from baseline quality of life at 6 months
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Get up from the chair 5 times test | Change from baseline result of the test at 6 months
  The Get up from your chair 5 times test is aimed at measuring the participant's functionality. It assesses the muscular power of the lower limbs during the exercise of getting up and sitting down from the chair.

SECONDARY OUTCOMES:
App Usability Questionnaire MAUQ | Up to 6 months
  MAUQ is a questionnaire that measures the usability of interactive medical mobile applications. It consists of 21 questions which are divided into three dimensions: the Ease of Use and Satisfaction dimension which covers items 1 to 8 and assesses the ease of use and user satisfaction of mHealth applications, the second dimension called System Information Structure which covers items 9 to 14 and refers to the information layout of the system and finally the third dimension Utility which contains the remaining items 15 to 21 and assesses the usefulness of the application. This questionnaire uses a seven-point seven-point Likert-type scale (1 = strongly disagree, 2 = disagree, 3 = somewhat disagree, 4 = neither disagree, 4 = neither disagree nor agree, 5 = somewhat agree, 6 = agree, and 7 = strongly disagree, 5 = somewhat agree, 6 = agree, and 7 = somewhat agree. 14 strongly agree)
App usage by users | Up to 12 months
  The metrics stored in the App server will allow to measure the usage of the app by users. Different metrics will be collected: number of app downloaded, number of registered users, number of active users, number of times the user has visit each module, the modules that received more visits, nº contents with more linkes.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Fullaondo Zabala, Principal Investigator — Biosistemak Institute for Health Systems Research
Locations (1):
- Irati, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Webpage of GATEKEEPER project — https://www.gatekeeper-project.eu/